CLINICAL TRIAL: NCT03658590
Title: Dexamethasone Effect on Induction Delivery Interval at Term Randomized Controlled Trial
Brief Title: Dexamethasone and Induction of Delivery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: samar sayed el sayed (Other)
Responsible Party: Sponsor-Investigator, samar sayed el sayed, Gynecologist and Obstetrician, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 100
Record Dates: First submitted 2018-08-29; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Induction of Labor Affected Fetus / Newborn
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group D (Active Comparator): including 51 women who will receive a prefilled syringe with two milliliters (8 mg) of dexamethasone intravenously.
  Interventions: Drug: Dexamethasone
- Group P (Placebo Comparator): including 51 women who will receive a prefilled syringe with two milliliters of distilled water intravenously.
  Interventions: Drug: Distilled Water

INTERVENTIONS:
Drug: Dexamethasone — a prefilled syringe with two milliliters (8 mg) of dexamethasone intravenously
  Other Names: Drug group
  Arms: Group D
Drug: Distilled Water — a prefilled syringe with two milliliters of distilled water intravenously.
  Other Names: Placebo group
  Arms: Group P

SUMMARY:
This study aims to evaluate the effect of intravenous injection of a single dose of dexamethasone in shortening the duration interval between initiation of labor induction and delivery of the fetus in primigravida full-term pregnancy.

DETAILED DESCRIPTION:
Research hypothesis:

In full term primigravidae undergoing induction of labor, the use of a single dose of dexamethasone (8mg) intra-venously will help in shortening the duration interval between initiation of labor induction and delivery of the fetus.

Research question:

In full term primigravidae undergoing induction of labor, does the use of intra-venous dexamethasone play a role in shortening the duration interval between initiation of labor induction and delivery of the fetus?

Patients and Methods

Type of study:

Double blind randomized controlled trial.

Study settings:

Site: Ain Shams Maternity Hospital Study duration: 6 months

Study population:

One hundred and two pregnant women will be recruited in this study from women attending the emergency room department of obstetrics and gynecology at Ain Shams University.

Inclusion criteria:

Primiparity Singleton pregnancy Gestational age i.e. 40 weeks or more by date or 1st trimestric ultrasound. Bishop score of 4 or greater. Longitudinal lie. Vertex presentation. Intact membranes

Exclusion criteria:

Refused consent Malpresentation. Multiple pregnancies. Active phase of labour. Rupture of membranes (ROM). Cephalo-pelvic disproportion. Previous C-section or myomectomy operation. Known contraindication or hypersensitivity to Dexamethasone. Fetal distress. IUFD Current maternal disorder e.g. diabetes mellitus and pregnancy induced hypertension.

Over distended abdomen e.g. fetal macrosomia or polyhydramonus suggested by ultrasound.

Ante-partum hemorrhage e.g. placenta previa, accidental hemorrhage.

These criteria will be assessed at first during the initial evaluation in the delivery suite as follows:

History:

Personal, menstrual, obstetric, past and family history will be taken. History of present pregnancy will be taken including the first day of last menstrual period, duration of pregnancy, warning symptoms as headache, visual symptoms, edema of face and fingers, excessive vomiting, heart burn, epigastric pain, vaginal bleeding, decreased fetal movements, edema of the lower limbs and history of any drug intake.

Examination:

1. General examination:vital signs, chest, heart and lower limb examination.
2. Abdominal examination: for assessment of fundal level, presentation, expected fetal weight, fetal heart rate and presence of scars of previous operations as cesarean section or myomectomy.
3. Vaginal examination: for assessment of cervical dilatation and effacement at the beginning, state of fetal membranes, station of fetal head, position of fetal head and pelvic adequacy.

Investigations:

1. Laboratory: blood grouping, Rh typing, complete blood count.
2. Abdominal ultrasound: to confirm the gestational age, fetal number, viability, presentation, position, estimated fetal weight, and to detect the grade of placental maturity, amount and turbidity of liquor.
3. CTG: application of CTG half an hour to all participates before starting any intervention.

Enrollment and Allocation of the patients:

After approval of health ethical committee in Ain Shams Hospital and after the initial evaluation, women who fulfilled the appropriate inclusion and exclusion criteria will be invited to participate in the study, a verbal consent will be obtained from each candidate after explanation of the procedure in details.

Randomization:

The eligible 102 women will be randomized into one of the following two groups:

1. Group D (study group): including 51 women who will receive a prefilled syringe with two milliliters (8 mg) of dexamethasone intravenously.
2. Group P (control group): including 51 women who will receive a prefilled syringe with two milliliters of distilled water intravenously.

No cervical ripping agent will be used for induction of labor in either group. Randomization is performed using a computer-generated randomization system. 102 opaque envelopes will be numbered serially; each envelope will contain the corresponding letter in the randomization table, and when the first pregnant woman arrived, the first envelope will be opened and the pregnant woman will be allocated to the group according to the inside letter.

ELIGIBILITY:
Inclusion Criteria:

* Primiparity
* Singleton pregnancy
* Gestational age i.e. 40 weeks or more by date or 1sttrimestric ultrasound.
* Bishop score of 4 or greater.
* Longitudinal lie.
* Vertex presentation.
* Intact membranes

Exclusion Criteria:

* Refused consent
* Malpresentation.
* Multiple pregnancies.
* Active phase of labour.
* Rupture of membranes (ROM).
* Cephalo-pelvic disproportion.
* Previous C-section or myomectomy operation.
* Known contraindication or hypersensitivity to Dexamethasone.
* Fetal distress.
* IUFD
* Current maternal disorder e.g. diabetes mellitus and pregnancy induced hypertension.
* Over distended abdomen e.g. fetal macrosomia or polyhydramonus suggested by ultrasound.
* Ante-partum hemorrhage e.g. placenta previa, accidental hemorrhage.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
The interval between the initiation of induction and the delivery of the fetus. | Up to 1 day
  Mean time of interval between the initiation of induction and the delivery of the fetus in the two groups.

SECONDARY OUTCOMES:
The duration of the first stage of labor (Partographic representation will do for each participant). | Up to 1 hour
  Mean time of duration of the first stage of labor in the two groups.
The duration of the second stage of labor. | Up to 2 hours
  Mean time of duration of the second stage of labor in the two groups.
The duration of the third stage of labor. | Up to 30 minutes
  Mean time of duration of the third stage of labor in the two groups.
The neonatal outcome by APGAR score. | at 1 and 5 minutes
  Mean of APGAR score at 1 and 5 minutes for fetus in the two groups.
Any postpartum maternal adverse effects (e.g. vital sing abnormality, any maternal postpartum hemorrhage and central nervous system manifestation). | Up to 1 day
  Percentage of postpartum adverse effects in both group.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek F Tamara, MD, Study Chair — Ain Shams University; Amgad E Abou Gamrah, MD, Study Director — Ain Shams University; Gihan E Elhawwary, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided